CLINICAL TRIAL: NCT04921449
Title: A Cluster-Randomized Trial of the Northwestern Embedded Emergency Department Physical Therapy (NEED-PT) Protocol for Acute Low Back Pain
Brief Title: ED Physical Therapy for Acute Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Howard Kim, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HS027426 (AHRQ)
Record Dates: First submitted 2021-05-18; First posted 2021-06-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Low Back Pain
Keywords: low back pain; physical therapy; emergency department; functioning; disability; opioid
MeSH Terms: conditions — Low Back Pain; Emergencies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Embedded ED Physical Therapy (NEED-PT) (Experimental): An ED physical therapist will be embedded with the primary treatment team to evaluate patients presenting with low back pain at the beginning of the overall treatment course. The physical therapist will utilize a clinical protocol (NEED-PT) that matches the patient's history and exam findings to an appropriate treatment classification consisting of directional preference exercises, manual traction, stabilization exercises, non-thrust manipulation/mobilization, and/or psychologically informed rehabilitation. The NEED-PT intervention will supplement any usual care performed by the treating physician.
  Interventions: Other: ED Physical Therapy
- Usual Care (Other): Usual care consists of any ED testing or treatment not involving an ED physical therapist in accordance with the treating physician's usual and customary practice. This could include diagnostic imaging, patient education and reassurance, and administration and/or prescribing of analgesic medications.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: ED Physical Therapy — All ED Physical Therapy treatment classifications involve a combination of exercise, range of motion, education, prognostic guidance, and reassurance. Patients are provided with an individualized home exercise plan based on their matched treatment classification and/or active rest.
  Arms: Embedded ED Physical Therapy (NEED-PT)
Other: Usual Care — Includes any diagnostic imaging, patient education and reassurance, and administration or prescribing of analgesic medications, as per the treating physician's usual and customary practice.
  Arms: Usual Care

SUMMARY:
Emergency department (ED)-initiated physical therapy is a rapidly growing resource and represents a promising treatment approach to low back pain. This clinical trial will evaluate an innovative model of an emergency department "embedded" physical therapist to treat patients with acute low back pain, with a focus on improving patient functioning and reducing opioid use.

DETAILED DESCRIPTION:
Low back pain represents a significant health care burden in the United States and accounts for nearly four million emergency department (ED) visits per year. In nearly two thirds of these visits, an opioid medication is administered or prescribed, making low back pain the most common reason for which opioids are prescribed. Despite this aggressive medication-based approach, patient outcomes after an ED visit for back pain remain poor: after three months, nearly half of all patients report persistent functional impairment, and one in five patients report continued opioid use.

ED-initiated physical therapy (ED-PT) is a promising new resource to improve patient care for low back pain. A growing number of EDs now have dedicated physical therapists that evaluate and treat patients through a combination of education, prognostic guidance, and early mobilization and exercise. Preliminary data indicate that patients receiving ED-PT, compared to usual care, report more rapid functional improvement and use fewer opioids. However, these observational data are limited by biases in treatment selection due to physician discretion in which patients receive ED-PT, as well as other measured and unmeasured confounders.

To more rigorously evaluate the efficacy of ED-PT for acute low back pain, the investigators will conduct a single-center physician-randomized trial of an embedded physical therapy intervention (NEED-PT) versus usual care in ED patients with acute low back pain, comparing a primary outcome of pain-related functioning and a secondary outcome of opioid use at the primary endpoint of three months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Low back pain (originating between 12th rib and buttocks)
* Symptom duration ≤ 30 days (current episode)
* Evaluated by a physician randomized to either study arm
* Evaluated when ED physical therapy is available (e.g., Mon-Fri, 8am-4pm)
* Likely to be discharged home (based on physician assessment)
* Ability to complete follow-up data collection electronically or by telephone
* English-speaking

Exclusion Criteria:

* Chronic low back pain or prior lumbar surgery
* Serious red-flag signs/symptoms (bladder/bowel incontinence, saddle anesthesia, debilitating motor weakness)
* Obvious non-musculoskeletal etiology for low back pain (e.g., shingles, kidney stone)
* Other concomitant injuries or pain (e.g., closed head injury, shoulder pain)
* Unable to ambulate at baseline
* Known pregnancy, under police custody, unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain Interference (PROMIS-PI) | Three months after the index ED visit.
  PROMIS-PI measures the self-reported consequences of pain on relevant aspects of a person's life, including social, cognitive, emotional, physical, and recreational activities. We will use the computer-adaptive format to minimize respondent burden. Scores are standardized to the general U.S. population, with a score of 50 representing the population mean. The time frame of interest for the PROMIS-PI is "in the past 7 days," meaning that participants provide responses based on their symptoms over the last week.

SECONDARY OUTCOMES:
Modified Oswestry Disability Index (ODI) | Three months after the index ED visit.
  The ODI contains 10 questions relating to low back pain intensity, personal care, lifting, walking, sitting, standing, sleeping, social life, traveling, and employment/homemaking. The ODI score ranges from zero (no disability) to 100 (maximum disability). The time frame of interest for the ODI is "today," meaning that participants provide responses based on their current symptoms on the day of survey response. The modified ODI replaces an item from the original ODI pertaining to sex life with a new item pertaining to employment/homemaking.
Patient-Reported Opioid Use in Last 24 Hours | Three months after the index ED visit.
  Patient-reported opioid use will be collected using a customized instrument assessing whether participants have taken any opioid medication in the last 24 hours (binary yes/no). The 24-hour timeframe was selected to maximize accuracy in patient recall and has been used previously. In brief, opioid medications are listed by brand and generic names; a "yes" response to any medication triggers an additional query asking the participant to specify the medication dose (e.g., oxycodone 10mg) and quantity (e.g., four pills), allowing for standardization by morphine milligram equivalents.

OTHER OUTCOMES:
Opioid Prescription Filling | Three months after the index ED visit.
  Opioid prescription filling data will be queried in the state prescription monitoring database.
Patient-Reported Prescription Analgesic Use in Last 24 Hours | Three months after the index ED visit.
  Patient-reported prescription analgesic use will be collected using the same customized instrument described above for opioid use. Prescription analgesics include the following: opioids, benzodiazepines, skeletal muscle relaxants, and gabapentinoids.
Prescription Analgesic Filling | Three months after the index ED visit.
  Prescription analgesic filling data will be queried in the state prescription drug monitoring database. Prescription analgesics include opioids, benzodiazepines, skeletal muscle relaxants, and gabapentinoids.
Numeric Pain Rating Scale (NPRS) | Three months after the index ED visit.
  The NPRS measures pain intensity from 0 to 10 and is easily understood by laypersons, clinicians, and researchers. We will assess a single item relating to average pain intensity over the last 24 hours.
Global Rating of Change (GROC) | Three months after the index ED visit.
  The GROC is a single-item survey used to evaluate overall recovery from low back pain from "the time that you began having pain until now." Responses are provided on a 15-point Likert scale ranging from "a very great deal worse" to "a very great deal better."
Pain Catastrophizing Scale (PCS-4) | Three months after the index ED visit.
  The original PCS is a 13-item survey measuring the degree to which an individual catastrophizes in response to pain. PCS scores correlate closely with pain intensity and disability over time; higher PCS scores are associated with progression from acute to chronic pain. We will utilize the brief 4-item PCS measure containing original items 3, 6, 8, and 11.
Pain Self-Efficacy Questionnaire (PSEQ-4) | Three months after the index ED visit.
  The original PSEQ is a 10-item survey measuring the confidence with which individuals can do things despite pain. We will utilize the brief 4-item PSEQ measure containing original items 4, 6, 8, and 9.
Advanced Healthcare Resource Utilization | Three months after the index ED visit.
  We will assess the proportion of participants who utilized any advanced healthcare resources for low back pain after their index ED visit, defined as advanced imaging (e.g., magnetic resonance imaging) or procedures/surgery (e.g., epidural steroid injection, lumbar discectomy).
ED Diagnostic Imaging Utilization | Index ED 1 day visit.
  We will assess the proportion of ED visits in which any diagnostic imaging of the lower back was performed, including plain radiography, computed tomography, or magnetic resonance imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Howard S Kim, MD MS, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) that underlie any published reports of this clinical trial (text, tables, figures, and appendices) will be made available upon reasonable request by qualified researchers engaging in independent scientific research and after review of the research proposal and execution of a data use authorization agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 12 months after article publication. Data will be made accessible for up to 12 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research. Access will be provided following review and approval of the research proposal and execution of data use authorization agreement.

REFERENCES:
- [Derived] Kim HS, Muschong KM, Fishman IL, Schauer JM, Seitz AL, Strickland KJ, Lambert BL, McCarthy DM, Vu MH, Ciolino JD. Embedded emergency department physical therapy versus usual care for acute low back pain: a protocol for the NEED-PT randomised trial. BMJ Open. 2022 May 24;12(5):e061283. doi: 10.1136/bmjopen-2022-061283. PMID 35613820

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04921449/SAP_001.pdf